CLINICAL TRIAL: NCT05297565
Title: A Phase 3, Open Label, Randomized, Non-Inferiority Pharmacokinetic Study of Nivolumab Subcutaneous (Nivo SC) Versus Intravenous (Nivo IV) Administration in Participants With Stage IIIA/B/C/D or Stage IV Adjuvant Melanoma Following Complete Resection
Brief Title: A Study to Compare Nivolumab Administered Subcutaneously vs Intravenous in Melanoma Participants Following Complete Resection
Acronym: CheckMate-6GE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-6GE; 2021-003208-42 (EudraCT Number); U1111-1266-6116 (Registry Identifier: WHO)
Expanded Access: NCT03126643 (Approved for marketing)
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Results first posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Melanoma
Keywords: Skin Cancer; rHuPH20; OPDIVO®
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Subcutaneous Nivolumab (Experimental)
  Interventions: Biological: Nivolumab/rHuPH20
- Arm B: Intravenous Nivolumab (Active Comparator)
  Interventions: Biological: Nivolumab

INTERVENTIONS:
Biological: Nivolumab/rHuPH20 — Specified dose on specified days
  Other Names: BMS-986298
  Arms: Arm A: Subcutaneous Nivolumab
Biological: Nivolumab — Specified dose on specified days
  Other Names: BMS-936558; Opdivo
  Arms: Arm B: Intravenous Nivolumab

SUMMARY:
The purpose of this study is to assess the safety and tolerability of subcutaneous nivolumab vs intravenous nivolumab in participants with completely resected Stage IIIA/B/C/D or Stage IV melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Stage IIIA/B/C/D or Stage IV melanoma and have histologically confirmed melanoma that is completely surgically resected (free of disease) with negative margins
* Complete resection performed within 12 weeks prior to randomization or treatment assignment
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1

Exclusion Criteria:

* History of uveal or mucosal melanoma
* Untreated/unresected CNS metastases or leptomeningeal metastases
* Active, known or suspected autoimmune disease
* Serious or uncontrolled medical disorder 4 weeks prior to screening
* Concurrent malignancy (present during screening) requiring treatment or history of prior malignancy active within 2 years prior to randomization or treatment assignment. Participants with history of prior early stage basal/squamous cell skin cancer or non-invasive or in situ cancers that have undergone definitive treatment at any time are eligible
* Prior immunotherapy treatments for any prior malignancies are not permitted

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (16):
- United States (2):
  - Local Institution - 0004, Fort Wayne, Indiana
  - Local Institution - 0044, Knoxville, Tennessee
- Australia (3):
  - Local Institution - 0038, Coffs Harbour, New South Wales
  - Local Institution - 0003, Wollongong, New South Wales
  - Local Institution - 0008, Bendigo, Victoria
- Local Institution - 0029, Ghent, Belgium
- Italy (2):
  - Local Institution - 0016, Milan
  - Local Institution - 0015, Napoli
- Poland (2):
  - Local Institution - 0034, Opole, Opole Voivodeship
  - Local Institution - 0036, Bydgoszcz
- Spain (5):
  - Local Institution - 0026, Barcelona
  - Local Institution - 0002, Madrid
  - Local Institution - 0043, Madrid
  - Local Institution - 0005, Seville
  - Local Institution - 0030, Valencia
- Local Institution - 0040, Leicester, Leicestershire, United Kingdom

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 14 participants were randomized and treated
Groups:
- Arm A: Nivo SC (BMS-986298) 600 mg with 8,000 U of rHuPH20 administered via 2 sequential injections Q2W. Nivo SC will be administered in-clinic through cycle 5, Day 1.
- Arm B: * Nivo IV (BMS-936558) 240 mg Q2W for Cycles 1 through 4.
  * Nivo IV 480 mg Q4W Cycle 5 onwards for up to total of 52 weeks.
  * All dosing will be performed in-clinic.
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 6 | 8
Completed | 5 | 6
Not Completed | 1 | 2
Not completed — Other Reasons | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Disease recurrence | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 7 | 12
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 8 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 8 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered study treatment that does not necessarily have a causal relationship with this treatment.
  An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Time Frame: From first dose to 100 days post last dose (Approximately up to 14 Months)
Population: All Treated Participants
Measure: Number; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 6 | 8
Participants
  Any Grade | 6 | 8
  Grade 3 to 4 | 0 | 2
  Grade 5 | 0 | 0

2. Primary Outcome: Number of Participants With Serious Adverse Events
Description: A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose:
  * Results in death.
  * Is life-threatening (defined as an event in which the participant was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe).
  * Requires inpatient hospitalization or causes prolongation of existing hospitalization.
Time Frame: From first dose to 100 days post last dose (Approximately up to 14 Months)
Population: All Treated Participants
Measure: Number; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 6 | 8
Participants
  Any Grade | 0 | 0
  Grade 3 to 4 | 0 | 0
  Grade 5 | 0 | 0

3. Primary Outcome: Number of Participants With Treatment Related Adverse Events
Description: An adverse event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered study treatment.
  An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom or disease.
Time Frame: From first dose to 100 days post last dose (Approximately up to 14 Months)
Population: All Treated Participants
Measure: Number; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 6 | 8
Participants
  Any Grade | 6 | 8
  Grade 3 to 4 | 0 | 2
  Grade 5 | 0 | 0

4. Primary Outcome: Number of Participants With Treatment Related Serious Adverse Events
Description: as for outcome 2
Time Frame: From first dose to 100 days post last dose (Approximately up to 14 Months)
Population: All Treated Participants
Measure: Number; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 6 | 8
Participants
  Any Grade | 0 | 0
  Grade 3 to 4 | 0 | 0
  Grade 5 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events: (From first dose to last dose + 100 days): Approximately 14 Months All-Cause mortality (From randomization to end of study): Approximately 14 Months
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Arm/Group | Arm A | Arm B
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 6/6 | 8/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=6) | Arm B (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Tongue pruritus (Gastrointestinal disorders) | 1 | 0
Administration site reaction (General disorders) | 1 | 0
Asthenia (General disorders) | 4 | 1
Device related thrombosis (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Impaired healing (General disorders) | 1 | 0
Injection site pain (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1
Puncture site erythema (General disorders) | 1 | 0
Puncture site inflammation (General disorders) | 1 | 0
Puncture site pain (General disorders) | 1 | 0
Puncture site pruritus (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Body tinea (Infections and infestations) | 1 | 0
Bronchiolitis (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Gastrointestinal viral infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 2
Nasopharyngitis (Infections and infestations) | 2 | 1
Oral herpes (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Lipase increased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 3
Insomnia (Psychiatric disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Menstrual disorder (Reproductive system and breast disorders) | 1 | 0
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema nummular (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2
Hypertension (Vascular disorders) | 0 | 4
Lymphoedema (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-25): https://cdn.clinicaltrials.gov/large-docs/65/NCT05297565/Prot_SAP_000.pdf